CLINICAL TRIAL: NCT06693960
Title: Evaluating the Pharmacokinetics of Oregano and Potential Oregano-drug Interactions Using a Drug Cocktail Approach
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Office of Dietary Supplements (ODS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20296; U54AT008909 (NIH)
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Interaction
Keywords: pharmacokinetics; drug interaction; natural products; oregano; cytochrome P450; cocktail

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: oregano alone (Experimental): 6 participants will be administered 180 mg of a well-characterized oregano product. Blood will be drawn via an indwelling venous catheter immediately before and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours after administration of oregano. Urine will be collected in multiple jugs for 24 hours.
  Interventions: Dietary Supplement: Oregano
- Arm 2: drug cocktail alone (Experimental): 16 participants, which may or may not include any number of the original 6 from Arm 1, will be administered an oral drug cocktail consisting of caffeine (100 mg), dextromethorphan (30 mg), losartan (25 mg), midazolam syrup (2 mg), and omeprazole (20 mg). Blood and urine will be collected in the same manner described in Arm 1.
  Interventions: Drug: Drug cocktail
- Arm 3: acute oregano + cocktail (Experimental): The same 16 participants will be administered the oregano product and the drug cocktail. Blood and urine will be collected in the same manner described in Arm 1.
  Interventions: Dietary Supplement: Oregano; Drug: Drug cocktail
- Arm 4: chronic oregano + cocktail (Experimental): The same 16 participants will self-administer the oregano product at home for 5 consecutive days. On day 6, participants will return to the study setting, where the procedure described in Arm 3 will be repeated.
  Interventions: Dietary Supplement: Oregano; Drug: Drug cocktail

INTERVENTIONS:
Dietary Supplement: Oregano — Oil of oregano administered as a softgel (180 mg).
  Arms: Arm 1: oregano alone; Arm 3: acute oregano + cocktail; Arm 4: chronic oregano + cocktail
Drug: Drug cocktail — Oral drug cocktail consisting of caffeine (100 mg), dextromethorphan (30 mg), losartan (25 mg), midazolam syrup (2 mg), and omeprazole (20 mg).
  Arms: Arm 2: drug cocktail alone; Arm 3: acute oregano + cocktail; Arm 4: chronic oregano + cocktail

SUMMARY:
The purpose of this clinical trial is to determine how the supplement oregano affects how the body metabolizes pharmaceutical drugs.

DETAILED DESCRIPTION:
Oregano (Origanum vulgare) is a flowering plant native to Europe. The fresh or dried leaves are commonly used as a cooking herb. Oregano oil extracts are also marketed as herbal supplements. O. vulgare ranked as the number 12 top-selling herbal supplement in the natural channel in 2022. Oregano supplements are consumed for myriad purported medicinal properties, including antimicrobial, antioxidant, and anti-inflammatory effects. Oregano contains multiple types of compounds, including phenols, terpenes, and terpenoids. Recent compelling in vitro data showed that an extract of O. vulgare activated the human pregnane X receptor (PXR) and aryl hydrocarbon receptor (AhR), which regulate the expression and activity of the prominent drug metabolizing enzymes cytochrome P450 (CYP) 3A4 and CYP1A2, respectively. PXR also regulates the expression and activity of several other CYPs (e.g., CYP2C9, CYP2C19), as well as transporters (e.g., the efflux transporter P-glycoprotein (P-gp)). The extent of activation of both receptors by O. vulgare rivaled that of St. John's wort, a well-known herbal supplement that induces CYP and P-gp activity in human participants. These investigators next evaluated the effects of O. vulgare on CYP3A4 and CYP1A2 activity in human hepatocytes. Again, the extent of induction by O. vulgare rivaled that of St. John's wort. Collectively, these observations suggest that oregano supplements could precipitate numerous interactions with pharmaceutical drugs.

The primary objective of the proposed study is to evaluate the potential for a well-characterized O. vulgare product to precipitate pharmacokinetic interactions with a "cocktail" of oral drugs that are substrates for multiple CYPs. The investigators and others have shown this validated cocktail (caffeine, dextromethorphan, losartan, midazolam, and omeprazole) to be safe to administer to healthy adult participants. The secondary objective is to determine the pharmacokinetics of the oregano supplement, which to date have not been rigorously characterized in humans. Results will be used to help inform healthcare practitioners and consumers about the safe use of this increasingly popular herbal supplement when consumed with certain pharmaceutical drugs.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-64 years old and healthy
* Not taking any medications (prescription and non-prescription) or dietary/herbal supplements that can interfere with study drug pharmacokinetics
* Willing to abstain from consuming dietary/herbal supplements and citrus juices for several weeks
* Willing to abstain from cannabis/marijuana, hemp, and THC- and CBD-containing products for several weeks
* Willing to abstain from consuming caffeinated beverages or other caffeine-containing products the evening before and the morning of the first day of each study arm
* Willing to abstain from consuming any alcoholic beverages for at least 1 day prior to any study day and during the study day
* Willing to use a secondary method of birth control that does not include the introduction or discontinuance of hormonal-based birth control (such as abstinence, copper IUD, or condoms). Specifically, regardless of the use hormonal-based birth control, a non-hormonal method should be used for the duration of the study and for three weeks following cessation of participation.
* Willing to abstain from consuming oregano (as a food additive or otherwise) for the duration of the study
* Geographically located within a 40-mile radius of Spokane and have the time to participate

Exclusion Criteria:

* Under 18 or over 64 years old
* Taking medications or dietary/herbal supplements that can interfere with study drug pharmacokinetics
* Have a major illness
* Taking medication/supplements for a mineral deficiency
* History of intolerance or allergy to oregano or any of the cocktail drugs (caffeine, dextromethorphan, losartan, midazolam, and omeprazole)
* Use of cannabis/marijuana, hemp, and CBD- and/or THC-containing products within the last month
* Currently using drugs or illicit substances for recreational purposes
* Pregnant or nursing
* Geographically located outside the 40-mile radius of Spokane and do not have the time to participate
* Cannot read and speak English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Midazolam Area under the plasma concentration vs. time curve (AUC) ratio | 0-24 hours
  Ratio of the area under the plasma concentration vs. time curve of midazolam in the presence to absence of oregano.

SECONDARY OUTCOMES:
Caffeine AUC ratio | 0-24 hours
  Area under the plasma concentration vs. time curve of caffeine in the presence to absence of oregano.
Caffeine maximum plasma concentration (Cmax) ratio | 0-24 hours
  Ratio of the maximum plasma concentration of caffeine in the presence to absence of oregano.
Caffeine half-life ratio | 0-24 hours
  Ratio of the half-life of caffeine in the presence to absence of oregano.
Dextromethorphan AUC ratio | 0-24 hours
  Area under the plasma concentration vs. time curve of dextromethorphan in the presence to absence of oregano.
Dextromethorphan Cmax ratio | 0-24 hours
  Ratio of the maximum plasma concentration of dextromethorphan in the presence to absence of oregano.
Dextromethorphan half-life ratio | 0-24 hours
  Ratio of the half-life of dextromethorphan in the presence to absence of oregano.
Losartan AUC ratio | 0-24 hours
  Ratio of the area under the plasma concentration vs. time curve of losartan in the presence to absence of oregano.
Losartan Cmax ratio | 0-24 hours
  Ratio of the maximum plasma concentration of losartan in the presence to absence of oregano.
Losartan half-life ratio | 0-24 hours
  Ratio of the half-life of losartan in the presence to absence of oregano.
Midazolam Cmax ratio | 0-24 hours
  Ratio of the maximum plasma concentration of midazolam in the presence to absence of oregano.
Midazolam half-life ratio | 0-24 hours
  Ratio of the half-life of midazolam in the presence to absence of oregano.
Omeprazole AUC ratio | 0-24 hours
  Area under the plasma concentration vs. time curve of omeprazole in the presence to absence of oregano.
Omeprazole Cmax ratio | 0-24 hours
  Ratio of the maximum plasma concentration of omeprazole in the presence to absence of oregano.
Omeprazole half-life ratio | 0-24 hours
  Ratio of the half-life of omeprazole in the presence to absence of oregano.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication